CLINICAL TRIAL: NCT04769089
Title: Effects of Pulsed Dye and CO2 Laser in Treatment of Hypertrophic Burn Scars.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Metis Foundation (Other)
Collaborators: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rodney Chan, Investigator, The Metis Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-10590
Record Dates: First submitted 2021-02-08; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Therapeutics; Lasers, Gas

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Pulse Dye Laser (Experimental): Treatment with PDL alone.
  Interventions: Procedure: Treatment with Pulse Dye Laser
- CO2 Laser (Experimental): Treatment with CO2 alone.
  Interventions: Procedure: Treatment with CO2 Laser
- Combination (Experimental): Treatment with both PDL and CO2 laser.
  Interventions: Procedure: Treatment with combination of pulse dye laser and CO2 laser.
- No treatment (Active Comparator): No laser treatment.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Treatment with Pulse Dye Laser — Pulse Dye laser treatment will be applied to one randomized area with the 10mm hand piece, duration of 0.45ms, and fluence of 5.25J/s.
  Arms: Pulse Dye Laser
Procedure: Treatment with CO2 Laser — CO2 laser treatment will be applied to one randomized area with the deep Fx hand piece, 300Hz, 15mJ, 15% density.
  Arms: CO2 Laser
Procedure: Treatment with combination of pulse dye laser and CO2 laser. — Pulse Dye laser and CO2 treatment will be applied to one randomized area. Pulse Dye will be applied with the 10mm hand piece, duration of 0.45ms, and fluence of 5.25J/s followed by the CO2 laser treatment with the deep Fx hand piece, 300Hz, 15mJ, 15% density.
  Arms: Combination
Other: Control — One area will be randomized to receive no laser treatment.
  Arms: No treatment

SUMMARY:
A prospective, double blind, randomized controlled human clinical trial will be conducted by enrolling patients referred for laser treatment from the USAISR burn clinic. Laser candidates will be asked to participate who have an area of extremity or truncal scar measuring approximately 6cmX6cm total, in one contiguous region. The study sites, will consist of four equally sized treatment areas (3cm x 3cm), will be randomized to be treated with PDL, CO2, a combination of CO2+PDL, and an untreated control for 6 treatments. The areas will be photographed prior to each treatment and at the final visit 4-6 months after the last treatment. Color, pliability and thickness will be measured using a colorimeter, cutometer and high frequency ultrasound respectively at each appointment. Additionally, the Patient Observer Scar Assessment Scale (POSAS) will be used to score the quality of the scar, using two trained, blinded observers. The patients will also be asked on a voluntary basis for a pre-trial and post-trial 3mm punch biopsy to evaluate for the presence of histological changes.

ELIGIBILITY:
Inclusion Criteria:

1. Must have at least four areas of burn scar located on the trunk or extremities measuring 3cm x 3cm and not previously treated with laser.
2. Timing: There has been a minimum of 1 month after burn closure
3. The subject is at least 18 years of age and not older than 65.
4. Able and willing to provide verbal and written consent.

Exclusion Criteria:

1. Active infection in experimental area
2. Use of isotretinoin (Accutane) in last six months
3. Life or limb-threatening injury/disease
4. Prior history of non-compliance with medical regimes
5. Active drug use/abuse
6. Active psychiatric illness except depression (unless being treated for suicidal intentions)
7. Pregnancy
8. Active cancer, or new diagnosis of cancer within the past 5 years, with the exception of basal cell carcinoma, melanoma and squamous cell carcinoma, as long as the subject is disease free at the time of enrollment.
9. Prior PDL or other laser treatment of the study area.
10. Patient unable to tolerate laser procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Effectiveness of laser treatments | 4-6 weeks post treatment
  Using the Patient and Observer Scar Assessment Scale (POSAS), evaluate the effectiveness of Pulse Dye Laser (PDL) and Carbon Dioxide (CO2) laser treatment on symptoms related to Hypertrophic Burn Scar (HBS)

SECONDARY OUTCOMES:
Improvement of symptoms | 4-6 weeks post treatment
  To longitudinally compare the change in symptoms by treatment modality between treatment sessions by assessment with the Patient and Observer Scar Assessment Scale (POSAS) measured for each patient and two observers (to increase score reliability) at each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Chan, MD, Principal Investigator — Metis Foundation
Locations (1):
- United States Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooper LE, Nuutila K, Kemp Bohan PM, Diaz V, Batchinsky M, Carlsson AH, Cancio LC, Chan RK. Analysis of the Utility of CO2 and Pulse-Dye Lasers Together and Separately in the Treatment of Hypertrophic Burn Scars. Ann Plast Surg. 2022 Aug 1;89(2):166-172. doi: 10.1097/SAP.0000000000003240. PMID 35943226